CLINICAL TRIAL: NCT06909552
Title: Use of an Educational Video to Improve Caregiver Knowledge, Adherence to Recommendations, and Outcomes in Children With Dysfunctional Voiding
Brief Title: Use of an Educational Video to Improve Adherence to Treatment in Voiding Dysfunction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-1255
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Dysfunctional Voiding
Keywords: dysfunctional voiding; educational video; treatment adherence; behavioral modification
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Masking Description: masking is not feasible as the use of a video will be known to both researcher and patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Video (Experimental): Participants will be exposed to a short 3-minute educational video following a visit with their urology provider.
  Interventions: Other: Educational Video on Voiding Dysfunction
- Control (No Intervention): Participants will not be exposed to an educational video; rather, they will receive standard of care education in clinic regarding behavioral treatment modalities at home.

INTERVENTIONS:
Other: Educational Video on Voiding Dysfunction — The educational video is a short 3-minute video which describes the condition in detail, at the level that a parent or child could understand without a medical background.
  Arms: Educational Video

SUMMARY:
This study aims to see whether an educational video on a common urinary dysfunction leads to improved parent and child perceived adherence to treatments recommendations.

DETAILED DESCRIPTION:
This study aims to explore whether the use of an educational video on voiding dysfunction, a common urinary dysfunction, leads to improve parents and child perceived adherence to behavioral treatment recommendations. Our main hypothesis explores whether there is improved perceived adherence, and whether this improved perceived adherence leads to better symptom outcomes in this condition.

We do so through randomizing patients to a control and intervention group, where the latter is exposed to the educational video, while the control group experiences standard of care visits/follow-ups. Data is collected through surveys pre and post exposure to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Parents and Caregivers of pediatric urology patients with a diagnosis of Dysfunctional voiding (minimum 100 participants)
* 5-18 years old, no younger than 5 and no older than 18 years old
* Potty-trained - fully independent with toileting, can complete every step of the process and can do so satisfactorily by themselves.

Exclusion Criteria:

* Children with Voiding dysfunctionDysfunctional voiders with medically complex conditions (neurogenic bladder, POTS, EDS, etc.)
* Parent's child is notNot a first-time patient (i.e. has been seen in the past for dysfunctional voiding)
* Child has severeSevere intellectual disability, developmental delay, or cognitive impairment.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Perceived Adherence | 4 weeks, 8 weeks.
  Participants will take the TAPQ perceived adherence assessment at time points 4 weeks and 8 weeks.

SECONDARY OUTCOMES:
Video Acceptability | 0 weeks.
  Immediately after watching the educational video, participants will be asked to complete a questionnaire on the acceptability of the video. this will occur at time frame 0 weeks (for intervention group).
Dysfunctional Voiding Scoring System | 0 weeks, 4 weeks, and 8 weeks.
  Participants will be asked to complete a DVSS survey at timepoints 0 weeks, 4 weeks, and 8 weeks. This DVSS survey will be used to assess symptom improvement throughout the study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
resource limitations

REFERENCES:
- [Background] Feldman AS, Bauer SB. Diagnosis and management of dysfunctional voiding. Curr Opin Pediatr. 2006 Apr;18(2):139-47. doi: 10.1097/01.mop.0000193289.64151.49. PMID 16601493
- [Background] Dyson PA, Beatty S, Matthews DR. An assessment of lifestyle video education for people newly diagnosed with type 2 diabetes. J Hum Nutr Diet. 2010 Aug;23(4):353-9. doi: 10.1111/j.1365-277X.2010.01077.x. Epub 2010 May 20. PMID 20497292